CLINICAL TRIAL: NCT05419882
Title: Study of Perioperative Plasma Levels of Endothelial Glycocalyx Markers in Patients Undergoing Colon Surgery.
Brief Title: Perioperative Plasma Levels of Glycocalyx Markers in Colon Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Nuria García del Olmo, Medical Doctor Specialist in General Surgery and Digestive System, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: FISABIO
Record Dates: First submitted 2022-05-30; First posted 2022-06-15 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Endothelial Dysfunction
Keywords: Glycocalix; Heparan-sulphate; Syndecan-1; Colorectal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal surgery patients: In patients undergoing colorectal surgery, blood samples will be collected at 5 times: preoperatively, and at 2, 6, 24 and 48 hours after finishing surgery, respectively.

SUMMARY:
The glycocalyx is a layer of macromolecules that covers the luminal surface of the endothelium, playing an important role in vascular homeostasis. Several studies have shown that in conditions of sepsis there is a degradation of the glycocalyx mediated by inflammatory mechanisms, releasing its components into the bloodstream. These glycocalyx fragments can be measured in blood plasma, showing a correlation between these markers and organ dysfunction, severity and mortality in sepsis situations. However, despite the great interest in glycocalyx biomarkers, their values in patients undergoing colorectal surgery are not well known. Therefore, verifying whether plasma levels of glycocalyx damage markers increase in the perioperative period of colorectal surgery is of great interest at the pathophysiological and clinical level, since the correlation of these markers with postoperative clinical evolution is unknown. In this study we want to determine the plasma levels of Heparan-sulphate and Syndecan-1, two of the most important constituents of the glycocalyx, and perform several measurements to form a "time course" of the plasma levels of these markers, in order to compare the different subgroups of patients undergoing colorectal surgery based on their clinical and surgical characteristics.

DETAILED DESCRIPTION:
BACKGROUND: The endothelial glycocalyx (EG) is a complex layer of macromolecules that lines the luminal surface of the vascular endothelium. This concept was proposed more than 70 years ago and its composition is well studied as detailed in two reviews (1, 2). However, its role in the mechanisms of endothelial protection and injury, and its subsequent clinical implications, have recently become evident. The EG consists of a variety of molecules, including glycoproteins and proteoglycans, that provide the basis for plasma-endothelial cell interaction. The structure of EG, although well characterized in vitro, is poorly defined in vivo because its composition changes dynamically by self-assembly and shear-dependent enzymatic degradation or detachment of its elements. Its major components are hyaluronic acid, proteoglycans (PG) such as syndecan-1, glycoproteins, plasma proteins and glycosaminoglycans (GAG), whose main component is Heparan Sulfate. The EG as a whole forms an endothelial surface layer that acts as a barrier to circulating cells and large molecules. Considerable prognostic-therapeutic promise lies in the emergence of the EG as a key mediator of endothelial dysfunction in pathogenic states, particularly with respect to vascular permeability and edema formation. Several studies have demonstrated the role of EG in plasma/interstitial fluid balance (3,4,5), mechano-transduction that couples intravascular pressure, and endothelial cell responses, i.e., biochemical signals, (6) to the inflammatory response cascade (7,8,9). EG damage affects a number of important endothelial cell functions leading to impaired mechano-transduction with changes in fluid passage (6,10), activation of coagulation pathways (11), leukocyte adhesion (7,11 ) and platelets (12) to the surface of endothelial cells, and leakage of fluid and plasma proteins into the interstitium (13,14), resulting in tissue edema (15). The specific pathophysiological triggers that lead to EG damage are still actively investigated and remain poorly understood. Nevertheless, EG protection appears to be a promising target in many clinical scenarios, especially since its degradation is closely associated with the pathophysiology of inflammation, capillary leak, and edema formation in various injuries and disease states; including ischemia/reperfusion, hypoxia, inflammation, trauma, hypervolemia, atherosclerosis, diabetes, and hypertension (16). In patients undergoing major abdominal surgery (including digestive, urological, gynecological or other surgery) there is very little information on the potential endothelial damage secondary to surgery (19). There are some reviews that have studied the damage of the EG in septic patients of medical and surgical origin (17, 18). However, in relation to digestive abdominal surgery, and specifically in colorectal surgery, only one study has been carried out, with only 18 patients undergoing colectomy (without mentioning the pathologies) and they are included with other patients of major abdominal surgery of the pancreas, liver, gynecology and urology (19).

EXPECTED RESULTS: In this study, it is expected that in the patients who underwent elective surgery, the markers of glycocalyx damage will increase their values in the postoperative laboratory tests compared to the values of the baseline (control) laboratory tests. It is equally expected that in patients undergoing urgent surgery, generally in clinical states of occlusion, perforation or sepsis, with activation of the inflammatory response, dehydration with decreased oncotic pressure and generation of tissue edema and third space, the markers of damage of glycocalyx are already elevated in the baseline analysis, with a maintenance or greater elevation of its values in the postoperative period. Likewise, a correlation would be expected between glycocalyx damage markers and other markers involved in the inflammatory response, such as leukocytes, C-reactive protein, procalcitonin, and lactate; as well as with associated patient comorbidities that lead to endothelial degeneration, such as high blood pressure, obesity, diabetes, atherosclerosis, etc. If the results of this study were as expected, glycocalyx damage markers (Heparan sulfate and Syndecan-1) could be used together with other inflammatory markers (C-reactive protein, procalcitonin, etc.) and be very useful in postoperative follow-up. of surgical patients, being able to anticipate possible postoperative complications. However, if elevations in glycocalyx markers were not observed in the perioperative period, it could be due to a lack of the number of Time-course determinations; that is to say, that an elevation of markers did occur, but we would not have detected it in the measurement times; or a larger study population might also be needed. In either case, the study could be completed in subsequent research projects.

OBJECTIVES:

Primary Objectives: To estimate the plasma levels of the 2 most representative markers of damage to the endothelial glycocalyx (Heparan-sulphate and Syndecan-1) in patients undergoing colorectal surgery during the perioperative period ("time-course").

Secondary Objectives:

* To analyze a possible correlation of the Syndecan-1 and Heparan-sulphate levels with other analytical parameters (C-reactive protein, procalcitonin, lactate, blood count, coagulation and basic biochemistry).
* To analyze the possible relationof glycocalyx damage markers with different parameters depending on the patient (age, sex and associated comorbidities) and the surgical intervention (surgical time, approach route, type of surgery…).
* To analyze the possible relation of endothelial glycocalyx damage markers with other clinical parameters that may indicate a possible post-operative complication.

DESIGN METHODOLOGY: It is a clinical, prospective, observational, and longitudinal study of single-centre groups (Hospital Lluís Alcanyís, Xàtiva). Always after the approval of the Research Ethics Committee of said Hospital.

STUDY POPULATION: The study population (value of n ) has been calculated on a population of 100 patients who will undergo surgery approximately a year. With a confidence level of 95% and a margin of error of 5%, a sample size of 80 patients has been calculated. Said 80 patients will be older than age, men and women, undergoing elective or emergency colorectal surgery (right hemicolectomy, extended right hemicolectomy, left hemicolectomy, sigmoidectomy, anterior resection of the rectum or abdominoperineal amputation).

SELECTION OF PATIENTS AND INFORMED CONSENT: Selection of patients and the drafting of the informed consent documents will be carried out in a reasoned manner as established in article 32 of the Helsinki Declaration and in article 58.2 of the Biomedical Research Law. It must be considered taking into account the Declaration of Helsinki of the World Medical Association in its latest revision. And according to its latest version of the Declaration of Helsinki of Fortaleza (Brazil) October 2013. Patients will be included in the study upon preoperative hospital admission, after verifying compliance with the inclusion criteria. To participate, the signature of the informed consent will be required.

ELIGIBILITY:
Inclusion Criteria:

* Signing of the informed consent document.
* Age equal to or greater than 18 years.
* American Society of Anesthesiologists (ASA) surgical risk ≤ III.
* Undergoing colorectal surgery

Exclusion Criteria:

* Age < 18 years old
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population (value of n) has been calculated on a population of 100 patients who will undergo surgery approximately one year. With a confidence level of 95% and a margin of error of 5%, a sample size of 80 patients has been calculated. These 80 patients will be older than 18 years old, men and women, undergoing elective or emergency colorectal surgery (right hemicolectomy, extended right hemicolectomy, left hemicolectomy, sigmoidectomy, anterior resection of the rectum or abdominoperineal amputation)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
To analyze plasma levels changes of heparan-sulphate and syndecan-1 in perioperative period of colorectal surgery | Blood samples will be collected in 5 times: preoperatively, at 2 hours after surgery, 6 hours after surgery, 24 hours after surgery and 48 hours after surgery.
  To analyze plasma levels changes of glycocalyx damage markers (Heparan-sulphate and Syndecan-1) at 5 times: preoperatively, 2 hours after surgery, 6 hours after surgery, 24 hours after surgery, and 48 hours after surgery, to perform a "time cours" of the plasma levels of this markers. This determinations will be made by ELISA technique.

SECONDARY OUTCOMES:
C-reactive Protein, procalcitonin, lactate, complete blood count, coagulation and basic biochemistry | Blood samples will be collected in 5 times: preoperatively, at 2 hours after surgery, 6 hours after surgery, 24 hours after surgery and 48 hours after surgery.
  To analyze the possible correlation of the levels of Heparan-sulphate and Syndecan-1, with other analytical parameters (C-reactive protein, procalcitonin, lactate, complete blood count, coagulation and basic biochemistry).
To analyze the possible relationship of glycocalyx damage markers with different parameters depending on the patient and the surgical intervention | Blood samples will be collected in 5 times: preoperatively, at 2 hours after surgery, 6 hours after surgery, 24 hours after surgery and 48 hours after surgery.
  To analyze the possible relationship of glycocalyx damage markers with different parameters depending on the patient (age, sex and associated comorbidities) and the surgical intervention (surgical time, approach route, type of surgery...).
To study other clinical parameters that may indicate a possible postoperative complication and its relationship with markers of endothelial glycocalyx damage. | Blood samples will be collected in 5 times: preoperatively, at 2 hours after surgery, 6 hours after surgery, 24 hours after surgery and 48 hours after surgery.
  study other clinical parameters that may indicate a possible postoperative complication (such as paralytic ileus, anastomotic leak, abdominal collections...) and its relationship with markers of endothelial glycocalyx damage.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria García del Olmo, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Nuria Garcia Del Olmo, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reitsma S, Slaaf DW, Vink H, van Zandvoort MA, oude Egbrink MG. The endothelial glycocalyx: composition, functions, and visualization. Pflugers Arch. 2007 Jun;454(3):345-59. doi: 10.1007/s00424-007-0212-8. Epub 2007 Jan 26. PMID 17256154
- [Result] Weinbaum S, Tarbell JM, Damiano ER. The structure and function of the endothelial glycocalyx layer. Annu Rev Biomed Eng. 2007;9:121-67. doi: 10.1146/annurev.bioeng.9.060906.151959. PMID 17373886
- [Result] Vink H, Duling BR. Capillary endothelial surface layer selectively reduces plasma solute distribution volume. Am J Physiol Heart Circ Physiol. 2000 Jan;278(1):H285-9. doi: 10.1152/ajpheart.2000.278.1.H285. PMID 10644610
- [Result] van den Berg BM, Vink H, Spaan JA. The endothelial glycocalyx protects against myocardial edema. Circ Res. 2003 Apr 4;92(6):592-4. doi: 10.1161/01.RES.0000065917.53950.75. Epub 2003 Mar 13. PMID 12637366
- [Result] van Haaren PM, VanBavel E, Vink H, Spaan JA. Charge modification of the endothelial surface layer modulates the permeability barrier of isolated rat mesenteric small arteries. Am J Physiol Heart Circ Physiol. 2005 Dec;289(6):H2503-7. doi: 10.1152/ajpheart.00587.2005. Epub 2005 Aug 12. PMID 16100247
- [Result] Mochizuki S, Vink H, Hiramatsu O, Kajita T, Shigeto F, Spaan JA, Kajiya F. Role of hyaluronic acid glycosaminoglycans in shear-induced endothelium-derived nitric oxide release. Am J Physiol Heart Circ Physiol. 2003 Aug;285(2):H722-6. doi: 10.1152/ajpheart.00691.2002. Epub 2003 May 1. PMID 12730059
- [Result] Constantinescu AA, Vink H, Spaan JA. Endothelial cell glycocalyx modulates immobilization of leukocytes at the endothelial surface. Arterioscler Thromb Vasc Biol. 2003 Sep 1;23(9):1541-7. doi: 10.1161/01.ATV.0000085630.24353.3D. Epub 2003 Jul 10. PMID 12855481
- [Result] Mulivor AW, Lipowsky HH. Inflammation- and ischemia-induced shedding of venular glycocalyx. Am J Physiol Heart Circ Physiol. 2004 May;286(5):H1672-80. doi: 10.1152/ajpheart.00832.2003. Epub 2004 Jan 2. PMID 14704229
- [Result] Lipowsky HH. The endothelial glycocalyx as a barrier to leukocyte adhesion and its mediation by extracellular proteases. Ann Biomed Eng. 2012 Apr;40(4):840-8. doi: 10.1007/s10439-011-0427-x. Epub 2011 Oct 8. PMID 21984514
- [Result] Thi MM, Tarbell JM, Weinbaum S, Spray DC. The role of the glycocalyx in reorganization of the actin cytoskeleton under fluid shear stress: a "bumper-car" model. Proc Natl Acad Sci U S A. 2004 Nov 23;101(47):16483-8. doi: 10.1073/pnas.0407474101. Epub 2004 Nov 15. PMID 15545600
- [Result] Henry CB, Duling BR. TNF-alpha increases entry of macromolecules into luminal endothelial cell glycocalyx. Am J Physiol Heart Circ Physiol. 2000 Dec;279(6):H2815-23. doi: 10.1152/ajpheart.2000.279.6.H2815. PMID 11087236
- [Result] Vink H, Constantinescu AA, Spaan JA. Oxidized lipoproteins degrade the endothelial surface layer : implications for platelet-endothelial cell adhesion. Circulation. 2000 Apr 4;101(13):1500-2. doi: 10.1161/01.cir.101.13.1500. PMID 10747340
- [Result] Adamson RH. Permeability of frog mesenteric capillaries after partial pronase digestion of the endothelial glycocalyx. J Physiol. 1990 Sep;428:1-13. doi: 10.1113/jphysiol.1990.sp018197. PMID 2231409
- [Result] Huxley VH, Williams DA. Role of a glycocalyx on coronary arteriole permeability to proteins: evidence from enzyme treatments. Am J Physiol Heart Circ Physiol. 2000 Apr;278(4):H1177-85. doi: 10.1152/ajpheart.2000.278.4.H1177. PMID 10749712
- [Result] VanTeeffelen JW, Dekker S, Fokkema DS, Siebes M, Vink H, Spaan JA. Hyaluronidase treatment of coronary glycocalyx increases reactive hyperemia but not adenosine hyperemia in dog hearts. Am J Physiol Heart Circ Physiol. 2005 Dec;289(6):H2508-13. doi: 10.1152/ajpheart.00446.2005. Epub 2005 Jul 22. PMID 16040715
- [Result] Becker BF, Chappell D, Bruegger D, Annecke T, Jacob M. Therapeutic strategies targeting the endothelial glycocalyx: acute deficits, but great potential. Cardiovasc Res. 2010 Jul 15;87(2):300-10. doi: 10.1093/cvr/cvq137. Epub 2010 May 11. PMID 20462866
- [Result] Uchimido R, Schmidt EP, Shapiro NI. The glycocalyx: a novel diagnostic and therapeutic target in sepsis. Crit Care. 2019 Jan 17;23(1):16. doi: 10.1186/s13054-018-2292-6. PMID 30654825
- [Result] Yanase F, Naorungroj T, Bellomo R. Glycocalyx damage biomarkers in healthy controls, abdominal surgery, and sepsis: a scoping review. Biomarkers. 2020 Sep;25(6):425-435. doi: 10.1080/1354750X.2020.1787518. Epub 2020 Jul 4. PMID 32597227
- [Result] Steppan J, Hofer S, Funke B, Brenner T, Henrich M, Martin E, Weitz J, Hofmann U, Weigand MA. Sepsis and major abdominal surgery lead to flaking of the endothelial glycocalix. J Surg Res. 2011 Jan;165(1):136-41. doi: 10.1016/j.jss.2009.04.034. Epub 2009 May 20. PMID 19560161

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05419882/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05419882/ICF_001.pdf